CLINICAL TRIAL: NCT03733782
Title: Increasing Enteral Protein Intake in Critically Ill Trauma and Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Grant E. O'Keefe, Professor, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002185
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Critical Illness; Malnutrition; Enteral Nutrition; Protein Supplementation
MeSH Terms: conditions — Critical Illness; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modular enteral protein - Prosource (Active Comparator): Subjects are patients admitted to the surgical intensive care unit and identified by one of the investigators as being appropriate for protein supplementation. Guidelines required that patients were: 1. Deemed ready to start enteral nutritional support by the attending physician within 72 hours of admission to the intensive care unit, 2. No contraindications to full enteral support, 3. No history of chronic liver disease, 4. Serum creatinine < 2.0 mg/dl.
  Interventions: Dietary Supplement: Modular enteral protein - Prosource
- Control group (No Intervention): The investigators used the electronic medical record to identify control subjects. These were patients admitted to the surgical intensive care unit who were in the ICU long enough to undergo testing of 24 hour urine nitrogen excretion from January to December 2016.8 As part of standard clinical practice, measurement of urine nitrogen excretion is performed in patients who are in the ICU and receiving nutritional support for more than one week.

INTERVENTIONS:
Dietary Supplement: Modular enteral protein - Prosource — Supplemental protein (2 gm/kg/day of Prosource; Medtrition, Lancaster, PA) was administered via the nasal/oral feeding tube in 60 - 180 ml bolus infusions 2 - 4 times per day, independently of the enteral formula received. That is, the daily target amount of protein was initially administered as the supplement boluses and only after the enteral formula infusion approached the target rate was the amount of supplement decreased. Supplemental protein was reduced by 50% once the patient received 75% of targeted caloric intake over the previous day (0700 - 0700). Once the patient reached the target caloric intake for 48 hours, the amount of supplemental protein was decreased in order that the total protein prescribed equaled 2 gm/kg/day.
  Arms: Modular enteral protein - Prosource

SUMMARY:
Published guidelines recommend at least 2 gm/kg/day of protein for critically ill surgical patients. It may not be possible to achieve this level of intake using polymeric enteral nutritional formula and protein or amino acid supplementation will be necessary. This was a retrospective cohort study in which the investigators reviewed critically ill trauma and surgical patients treated with supplemental enteral protein according to a protocol aimed to deliver a total of 2 gm/kg/day of protein. The investigators studied detailed nutritional data from a 2 week period after admission and obtained additional data through discharge to determine caloric intake, protein intake and complications. The investigators also compared urine nitrogen excretion and visceral protein (transthyretin) concentrations between those who received early supplementation with those who did not.

DETAILED DESCRIPTION:
This is a retrospective analysis of a treatment approach designed to increase enteral protein intake in critically ill surgical patients. The study investigators recently developed guidelines aimed to improve early enteral protein delivery in critically ill patients. The guidelines were tested for 6 months; applying it to 53 patients (April to September, 2016) in order to determine its safety and effectiveness. All subjects were admitted to the surgical intensive care unit and identified by one of the investigators as being appropriate for protein supplementation. The guidelines required that patients were: 1. Deemed ready to start enteral nutritional support by the attending intensivist within 72 hours of admission to the intensive care unit, 2. No contraindications to full enteral support, 3. No history of chronic liver disease, 4. Serum creatinine <2.0 mg/dl.

In order to compare biochemical markers of nutritional support, the investigators used the electronic medical record to identify all patients admitted to the surgical intensive care unit who were in the ICU long enough to undergo testing of 24 hour urine nitrogen excretion from January to December 2016.8 As part of standard clinical practice, measurement of urine nitrogen excretion is performed in patients who are in the ICU and receiving nutritional support for more than one week. In addition to measuring TUN, the investigators also monitor the response to nutritional support and recovery from critical illness using serum transthyretin (also known as prealbumin).

This review resulted in a cohort of 118 patients who underwent at least one TUN measurement. Of these, 27 received early protein supplementation and 91 did not and these provide the basis for the comparisons described below. We wanted to measure the effect of early supplemental protein treatment on nitrogen excretion and on serum transthyretin concentrations as the patients recovered. We therefore, compared nitrogen excretion and serum transthyretin between those who received early supplementation and those who did not.

ELIGIBILITY:
Inclusion Criteria:

* All critically ill adult trauma (blunt and penetrating) and all surgical critical care patients ≥ 18 years old patients where enteral nutrition is begun by the attending physician during the first 48 hours after injury, and are expected to require nutritional support for at least 1 week

Exclusion Criteria:

* Significant chronic organ failure
* Severe malnutrition pre-existing prior to ICU admission
* Not expected to survive due to the severity of their illness or traumatic injuries
* Intestinal discontinuity
* Short bowel syndrome
* Bowel obstruction
* Enterocutaneous fistula
* Intestinal ischemia
* Massive gastrointestinal hemorrhage
* Inability to obtain enteral access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Enteral protein intake | 14 days
  Amount of enteral protein intake during first 14 days
Total urine nitrogen excretion | up to 2 weeks after admission
  Nitrogen excreted in urine over 24 hour period

SECONDARY OUTCOMES:
Ventilator-free days | Up to 28 days
  Days alive and not receiving mechanical ventilation in initial 28 days